CLINICAL TRIAL: NCT03826654
Title: Formulation of Vitamin D-fortified Sunflower Oil and Evaluation of the Efficacy of Its Consumption in Healthy Adults: a Randomized Controlled Clinical Trial
Brief Title: Assessment of the Efficacy of Vitamin D-fortified Oil in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, Ph.D., Prof., National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 24
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: vitamin D; fortified oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fortified oil (Experimental): daily intake of fortified sunflower oil (700IU vitamin D/ 35g)
  Interventions: Dietary Supplement: fortified oil
- control (Placebo Comparator): daily intake of plain oil
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fortified oil — 35 g fortified sunflower oil
  Arms: fortified oil
Dietary Supplement: Placebo — plain oil
  Arms: control

SUMMARY:
The aim of this study is to evaluate the efficacy of daily intake of fortified sunflower oil with vitamin D on serum 25-hydroxyvitamin D level, glycemic and lipidemic status in healthy subjects compared to plain oil.

DETAILED DESCRIPTION:
Sixty apparently healthy subjects will be selected. Participants who are receiving vitamin D, calcium or omega-3 supplements within the last three months will be excluded. Subjects will be assigned randomly to one of the two intervention groups: 1.fortified sunflower oil, 2. plain bread+vitamin D supplements,3. plain bread+placebo. Each participant will consume 50 g of oil every day for 2 months.

At the first and last visits, dietary and laboratory assessments will be performed for all subjects. Primary outcomes are the improvement in vitamin D status and secondary outcome is the improvement of glycemic and lipidemic markers and prevention of problems related to hypovitaminosis D.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 60 years
* healthy subjects
* no receiving vitamin D or omega-3 supplement in past 3 months

Exclusion Criteria:

- receiving vitamin D or omega-3 supplement during the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D (nmol/L) | 8 weeks

SECONDARY OUTCOMES:
serum glucose (mg/dL) | 8 weeks
serum triglyceride (mg/dL) | 8 weeks
serum total cholesterol (mg/dL) | 8 weeks
serum LDL | 8 weeks
serum HDL | 8 weeks
serum PTH (pg/mL) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, PhD, Study Chair — Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nikooyeh B, Zargaraan A, Kalayi A, Shariatzadeh N, Zahedirad M, Jamali A, Khazraie M, Hollis B, Neyestani TR. Vitamin D-fortified cooking oil is an effective way to improve vitamin D status: an institutional efficacy trial. Eur J Nutr. 2020 Sep;59(6):2547-2555. doi: 10.1007/s00394-019-02103-4. Epub 2019 Oct 12. PMID 31606753